CLINICAL TRIAL: NCT04717583
Title: Efficacy of Intense Pulsed Light (IPL) in the Treatment of Facial Telangiectasia in Patients With Systemic Lupus Erythematosus (SLE): a Randomized, Evaluator-blinded, Split-face Comparative Clinical Trial
Brief Title: Efficacy of Intense Pulsed Light in the Treatment of Facial Telangiectasia in Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Qianjin Lu, MD, PhD, Professor and Director, Institute of Dermatology, The Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SecondXHCSU-PFK2020SLE01
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Facial Telangiectasia in Patients With Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Intense pulsed light; Facial telangiectasia; corticosteroids
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPL-treated side (Experimental): For each participant, the two sides of face will be randomized into an IPL-treated side and a control side. In the first 3 visits, the IPL-treated side of the face will be treated with IPL, once every 4 weeks for 3 consecutive times.
  Interventions: Procedure: Intense pulsed light (IPL) treatment
- Control side (No Intervention): For each participant, the two sides of face will be randomized into an IPL-treated side and a control side. In the first 3 visits (before Week 12), the control side of face will not be treated by IPL.
  Starting from Week 12 (the time point of the primary endpoint), the control side of face will also be treated by IPL if the IPL-treated side shows satisfactory improvement of erythema or telangiectasia by IPL treatment. If the patient was unsatisfied with the improvement in the IPL-treated side at Week 12 visit, no IPL treatment will be given to either side of the face any more.

INTERVENTIONS:
Procedure: Intense pulsed light (IPL) treatment — After randomization, one side of the face will be treated with IPL using the M22™ Universal IPL device, once every 4 weeks for 3 consecutive times.
  Starting from Week 12 (the time point of the primary endpoint), the control side of face will also be treated by IPL if the IPL-treated side shows satisfactory improvement of erythema or telangiectasia by IPL treatment. If the patient was unsatisfied with the improvement in the IPL-treated side at Week 12 visit, no IPL treatment will be given to either side of the face any more.
  Arms: IPL-treated side

SUMMARY:
This clinical trial intends to evaluate the efficacy and safety of intense pulsed light (IPL) in the treatment of facial telangiectasia in patients with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease that can involve multiple organs and systems. The treatment for SLE mainly depends on long-term use of glucocorticoids. For many patients with SLE, facial telangiectasia is a commonly seen side effect of long-term use of glucocorticoids. Featured by facial erythema with or without flushing or burning sensation, facial telangiectasia seriously affects the quality of life of patients. However, up to now, there has been little attention paid to this condition in SLE patients. There have been a lack of effective treatment options for tackling this problem.

Intense pulsed light (IPL) is a non-laser light source used to treat a variety of vascular and pigmented lesions. Unlike ultraviolet that is harmful to patients with SLE, application of IPL may be a safe and effective treatment for SLE patients with facial telangiectasia. This study intends to evaluate the efficacy and safety of IPL in the treatment of facial telangiectasia for SLE patients that has been treated with long-term corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: between 18 and 65 years; 2. Patients definitedly diagnosed with systemic lupus erythematosus according to "Diagnostic Criteria for systemic lupus erythematosus"; 3. Patients receiving continuous treatment of glucocorticoid in the last 4 weeks.

Exclusion Criteria:

* 1. Patients with severe diseases of heart, brain, lungs, liver, kidney, or blood system; 2. Patients with drug abuse, alcohol abuse, or mental disorders that are unable to cooperate or adhere to treatment; 3. Pregnant women, lactating women or women who are ready to conceive within 6 months; 4. Participated in other clinical trials within 3 months before the screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change of Five-Point Telangiectasia Scale after three times of IPL treatment | 12 weeks
  Five-Point Telangiectasia Scale will be used to assess improvement of telangiectasia and erythema. The range of TGS is 1 to 5, where 1 means less than 5% clearance, 2 means 5-25% clearance, 3 means 25-50% clearance, 4 means 50-75% clearance, and 5 means 75-100% clearance, compared to baseline before IPL treatment.

SECONDARY OUTCOMES:
Change of Five-Point Telangiectasia Scale after 4, 8, and 24 weeks, respectively. | 4, 8, and 24 weeks
  Five-Point Telangiectasia Scale will be used to assess improvement of telangiectasia and erythema. The range of TGS is 1 to 5, where 1 means less than 5% clearance, 2 means 5-25% clearance, 3 means 25-50% clearance, 4 means 50-75% clearance, and 5 means 75-100% clearance, compared to baseline before IPL treatment.
Change of Clinician's Erythema Assessment (CEA) scores after a 4-, 8-, 12- and 24-week treatment, respectively. | 4, 8, 12, and 24 weeks
  Clinician's Erythema Assessment (CEA) scores describe the severity of facial erythema, ranging from 0-4. In CEA scoring system, 0=clear, and 4=severe.
Change of Patient Global Assessment (PGA) after a 4-, 8-, 12- and 24-week treatment, respectively. | 4, 8, 12, and 24 weeks
  PGA refers to the subject's global assessment of the facial telangiectasia condition. Change of PGA from baseline to post-treatment will be determined.
Change of Dermatology Life Quality Index (DLQI) scores after a 4-, 8-, 12-, and 24-week of treatment, respectively. | 4, 8, 12, and 24 weeks
  Change of DLQI from baseline to post-treatment will be determined.
Change of Skindex-16 scores after a 4-, 8-, 12- and 24-week of treatment, respectively. | 4, 8, 12, and 24 weeks
  Change of Skindex-16 from baseline to post-treatment will be determined.
The safety evaluation about the adverse reactions throughout the entire study process. | 4, 8, 12, 16, and 36 weeks
  The possible adverse reactions of IPL include rash, pain, short-term pigmentation, recurrence of telangitic erythema, recurrence or aggravation of SLE
Change of SLEDAI scores after 12 and 24 weeks, respectively | 12 and 24 weeks
  SLEDAI reflects the disease activity of SLE. A dramatic increase of SLEDAI during the IPL treatment or immediately after IPL treatment will be considered as an adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Human, China

IPD SHARING:
Plan to Share IPD: No